CLINICAL TRIAL: NCT03491527
Title: Influence of Resin Cement Composition on the Longevity of Intraradicular Post in the Rehabilitation of Endodontically Treated Teeth - Randomized Clinical Trials
Brief Title: Influence of Resin Cement Composition on the Longevity of Intraradicular Post of Endodontically Treated Teeth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Federal University of Uberlandia (Other)
Responsible Party: Principal Investigator, PAULO VINICIUS SOARES, Director of NCCL Research Group, Federal University of Uberlandia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2.570.182
Record Dates: First submitted 2018-04-02; First posted 2018-04-09 (Actual); Last update posted 2018-04-09 (Actual); Status verified 2018-04

CONDITIONS: MTA; Endodontically Treated Teeth; Resin Cement
MeSH Terms: conditions — Tooth, Nonvital | interventions — Pemetrexed; Dental Impression Technique; Occlusal Adjustment

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Resin Cement (Active Comparator): Resin cement without MTA
  Interventions: Procedure: Absolute isolation; Procedure: Manipulation of the resin cement without MTA; Procedure: Fiber Post cimentation; Procedure: Dental Prepare; Procedure: Dental impression; Procedure: Crown cimentation; Procedure: Occlusal adjustment
- MTA Resin Cement (Active Comparator): Resin cement with MTA
  Interventions: Procedure: Absolute isolation; Procedure: Manipulation of the resin cement with MTA; Procedure: Fiber Post cimentation; Procedure: Dental Prepare; Procedure: Dental impression; Procedure: Crown cimentation; Procedure: Occlusal adjustment

INTERVENTIONS:
Procedure: Absolute isolation — Absolute isolation with rubber dam
Procedure: Manipulation of the resin cement with MTA — Manipulation of the resin cement with MTA according to the manufacturer's recommendations.
  Arms: MTA Resin Cement
Procedure: Manipulation of the resin cement without MTA — Manipulation of the resin cement without MTA according to the manufacturer's recommendations.
  Arms: Conventional Resin Cement
Procedure: Fiber Post cimentation — Insertion of the cement on the root canal and on post surface. Light-cured for 40 seconds on each surface.
Procedure: Dental Prepare — Confection of a indirect crown prepare with diamand burs.
Procedure: Dental impression — Dental impression whith silicone.
Procedure: Crown cimentation — Insertion of the cement on the inner surface of the crown. Light-cured for 40 seconds on each surface.
Procedure: Occlusal adjustment — Analysis of the occlusion with carbon paper.

SUMMARY:
The aim of this study is through a randomized clinical trial, double blind, splithmouth, evaluate the success rate (post or dental crown displacement; fracture of the core/post/crown; marginal integrity and absence of endotontic alterations) of definitive indirect crowns un endodontically treated teeth. The composition of the resin cement (with and without mineral trioxide aggregate) will be evaluated. Data will be collected, tabulated and submitted to statistical analysis.

DETAILED DESCRIPTION:
Endodontically treated teeth present an increased risk of fracture and are usually related to extensive carious processes or trauma that promote major coronary destruction. In such situations, it may be necessary to indicate intra-radicular retainers, such as fiberglass pins, to retain the restorative material. The aim of this study is through a randomized clinical trial, double blind, splithmouth, evaluate the success rate (post or dental crown displacement; fracture of the core/post/crown; marginal integrity and absence of endotontic alterations) of definitive indirect crowns un endodontically treated teeth. The composition of the resin cement (with and without mineral trioxide aggregate) will be evaluated. Twenty participants with at least two teeth with endodontic treatment with need intraradicular post cementation and confection of indirect dental crown (each participant) will be selected. The teeth will be randomly divided into 2 different groups according to resin cement composition (with and without mineral trioxide aggregate). Data will be collected, tabulated and submitted to statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers;
* Presence of at least two teeth with endodontc treatment;
* Presence of at least two teeth with indication of total crowns;
* Good oral hygiene.

Exclusion Criteria:

* Dentures or orthodontics;
* Presence of periodontal disease
* Presence of parafunctional habits
* Presence of systemic disease
* Constant use of analgesic and or anti-inflammatory
* Allergic response to dental products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-05-01 (Estimated); Primary Completion 2018-09-30 (Estimated); Study Completion 2019-07-30 (Estimated)

PRIMARY OUTCOMES:
Success rate (post or dental crown displacement; fracture of the core/post/crown; marginal integrity and absence of endotontic alterations) of definitive indirect crowns with a 1 year follow up. | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Uberlandia, Uberlândia, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Assif D, Gorfil C. Biomechanical considerations in restoring endodontically treated teeth. J Prosthet Dent. 1994 Jun;71(6):565-7. doi: 10.1016/0022-3913(94)90438-3. PMID 8040817
- [Background] Bahari M, Savadi Oskoee S, Kimyai S, Mohammadi N, Saati Khosroshahi E. Effect of Light Intensity on the Degree of Conversion of Dual-cured Resin Cement at Different Depths with the use of Translucent Fiber Posts. J Dent (Tehran). 2014 May;11(3):248-55. Epub 2014 May 31. PMID 25628659
- [Background] Camilleri J, Montesin FE, Brady K, Sweeney R, Curtis RV, Ford TR. The constitution of mineral trioxide aggregate. Dent Mater. 2005 Apr;21(4):297-303. doi: 10.1016/j.dental.2004.05.010. PMID 15766576
- [Background] Christensen GJ. Post concepts are changing. J Am Dent Assoc. 2004 Sep;135(9):1308-10. doi: 10.14219/jada.archive.2004.0406. PMID 15493395
- [Background] Duarte MA, De Oliveira Demarchi AC, Yamashita JC, Kuga MC, De Campos Fraga S. Arsenic release provided by MTA and Portland cement. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2005 May;99(5):648-50. doi: 10.1016/j.tripleo.2004.09.015. PMID 15829892
- [Background] Lee SJ, Monsef M, Torabinejad M. Sealing ability of a mineral trioxide aggregate for repair of lateral root perforations. J Endod. 1993 Nov;19(11):541-4. doi: 10.1016/S0099-2399(06)81282-3. PMID 8151240
- [Background] Santos-Filho PC, Castro CG, Silva GR, Campos RE, Soares CJ. Effects of post system and length on the strain and fracture resistance of root filled bovine teeth. Int Endod J. 2008 Jun;41(6):493-501. doi: 10.1111/j.1365-2591.2008.01383.x. Epub 2008 Apr 12. PMID 18422584
- [Background] von Arx T. [Mineral trioxide aggregate (MTA) a success story in apical surgery]. Swiss Dent J. 2016;126(6):573-95. doi: 10.61872/sdj-2016-06-02. French, German. PMID 27377433